CLINICAL TRIAL: NCT05008601
Title: Detection of Cardiac Arrhythmias With Wrist-worn Combined Optical and ECG Based Heart Rate Monitor During Normal Daily Living
Brief Title: Aino ECG Ambulatory Study
Status: Completed | Type: Observational
Sponsor: PulseOn Oy (Industry)
Collaborators: TAYS Sydänkeskus Oy (Unknown); Atostek Oy (Unknown)
Responsible Party: Sponsor
Other Study IDs: AinoECG_Ambulatory
Record Dates: First submitted 2021-07-30; First posted 2021-08-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-08

CONDITIONS: Arrhythmias, Cardiac; Atrial Fibrillation and Flutter
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wrist-word optical heart rate and ECG measurement device — Aino ECG: wrist-word optical heart rate and ECG measurement device

SUMMARY:
The study includes collection of data from patients referred to a therapeutic evaluation in Tays Sydänkeskus Oy (Heart Center Co, Tampere University Hospital) or another unit of Sydänkeskus (hereafter the Heart Hospital) due to suspected cardiac arrhythmia. Data collection takes place outside the hospital in normal daily conditions. The monitoring is started during the outpatient visit at Heart hospital polyclinic or when leaving home from cardiac ward and it continues for 2 days. Reference information about the occurrence of arrhythmia episodes and the reference ECG data are obtained from simultaneously worn Holter device.

During the two days the study device and the reference device are worn continuously. Wearing the devices does not affect the daily routines of the participant except there is no possibility to take a shower. The arrhythmia episodes are labelled in post-hoc signal analysis and annotations visually confirmed by a cardiologist. The participants are instructed to take ECG recordings with the wrist device every time the device gives a notification and also whenever the participant feels arrhythmia symptoms. There will be at least four intermittent ECG records taken on each day.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* Suspected or earlier diagnosed episodic cardiac arrhythmia, for example atrial fibrillation or atrial flutter
* Ability to give informed consent
* Volunteering for the study

Exclusion Criteria:

* Implanted permanent pacemaker
* Inability to give informed consent e.g. due to mental confusion
* Denial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population of the study includes patients referred to a therapeutic evaluation or treatment in Tays Heart Hospital due to suspected cardiac arrhythmia. A portion (up to one third) of the subjects may be having on-going atrial fibrillation at the beginning of the measurement and may suffer from persistent or permanent atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Verification that the atrial fibrillation detection sensitivity satisfies the design input requirements defined for the Aino ECG device | 6 months
Verification that the data accuracy (accuracy of optically measured inter-beat-intervals) satisfies the design input requirement defined for the Aino ECG device. | 6 months
Verification that the quality of the ECG signal measured with Aino ECG satisfies the design input requirement defined for the Aino ECG device. | 6 months

SECONDARY OUTCOMES:
Showing that the quality of the measured PPG signal is similar enough compared with the one measured with the earlier prototype | 6 months
To obtain feedback regarding the usability of the Aino ECG wrist device | 6 months
  The feedback is obtained with feedback form filled by the study participants. The form includes questions regarding: overall impression on the study device, easiness of noticing and interpret the notifications of the device, comfortability of using the device, easiness of adjusting the tightness of the wrist band, and operation of the intermittent ECG measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Hernesniemi, Docent, Principal Investigator — Tampere Heart Hospital
Locations (1):
- Tampere Heart Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saarinen HJ, Joutsen A, Korpi K, Halkola T, Nurmi M, Hernesniemi J, Vehkaoja A. Wrist-worn device combining PPG and ECG can be reliably used for atrial fibrillation detection in an outpatient setting. Front Cardiovasc Med. 2023 Feb 9;10:1100127. doi: 10.3389/fcvm.2023.1100127. eCollection 2023. PMID 36844740